CLINICAL TRIAL: NCT06423521
Title: Value Analysis in Patients Undergoing Anticoagulant Therapy: Impact of Self-management Training Using a Coagulometer
Brief Title: Value Analysis in Patients Undergoing Self-Management Training Using a Coagulometer
Acronym: VAPUST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ana Rita Londral, PhD (Other)
Collaborators: NOVA Medical School (Other); Roche Diagnostics GmbH (Industry)
Responsible Party: Sponsor-Investigator, Ana Rita Londral, PhD, Director, Value for Health CoLAB
Organization: Value for Health CoLAB (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 1057/2021
Record Dates: First submitted 2024-05-15; First posted 2024-05-21 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Post-Cardiac Surgery Patients
Keywords: Digital healthcare; Telemedice; Remote Patient Monitoring; Antocoagulation Therapy
MeSH Terms: interventions — Standard of Care; Remote Patient Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SOC-RPM (Experimental): SOC-RPM arm, would follow the Standard of Care (SOC) for the first six months and then receive the Remote Patient Monitoring (RPM).
  Interventions: Other: Standard of Care (SOC)
- RPM-SOC (Experimental): RPM-SOC arm: would receive the intervention (RPM) for the first six months and then follow the SOC for the remaining six months.
  Interventions: Other: Remote Patient Monitoring (RPM)

INTERVENTIONS:
Other: Standard of Care (SOC) — The SOC intervention constitutes the common clinical practice of care that is habitually performed after cardiac surgery to manage anticoagulation therapies.
  Arms: SOC-RPM
Other: Remote Patient Monitoring (RPM) — The RPM intervention involves the use of a remote patient monitoring (RPM) system with a portable coagulometer for the clinical follow-up and self-management of International Normalized Ratio (INR) control in patients undergoing anticoagulant therapy post-cardiac surgery. Patients were provided with a Coagulometer-CoaguChek® (Roche Diagnostics, Switzerland) kit and test strips, along with written instructions for conducting measurements. They were also enrolled in a monitoring platform. Patients received regular text messages on their smartphones to report their INR values and symptoms related to anticoagulant therapy. The clinical team received notifications if patients' reports fell outside therapeutic standards and then responded with medication adjustments via text message.
  Arms: RPM-SOC

SUMMARY:
Prior research has not assessed the value of remote patient monitoring (RPM) systems for patients undergoing anticoagulation therapy after cardiac surgery. This study aims to assess whether the clinical follow-up through RPM yields comparable outcomes with the standard protocol. A crossover trial assigned participants to SOC-RPM or RPM-SOC, starting with the standard of care (SOC) for the first 6 months after surgery and using RPM for the following 6 months, or vice-versa, respectively. During RPM, patients used the Coaguchek© to accurately measure International Normalized Ratio values and a mobile text-based chatbot to report PROs and adjust the therapeutic dosage. The study assessed patients' and clinicians' experience with RPM and compared direct costs.

DETAILED DESCRIPTION:
The main objective of this pilot study was to evaluate the outcomes and costs of a digital clinical service to support patients with anticoagulant therapy after cardiac surgery. This study used an RPM-based system with a portable coagulometer for clinical follow-up and self-management of INR control and compared with the standard of care (SOC). In addition, this study seeks to assess patients' and clinical teams' satisfaction and experience.

Patients were recruited in sequential order based on their availability in the cardiothoracic surgery department. The participants were assigned into two arms: one would follow the SOC for the first six months and then receive the RPM intervention for the following six months (SOC-RPM); the other group would receive the intervention (RPM) for the first six months and then follow the SOC for the remaining six months (RPM-SOC). Blinding was not feasible due to the nature of the trial, and both patients and the clinical team were aware of the follow-up being conducted. In this study, it was decided that a washout period was not required. This was because withdrawing effective follow-up care for a washout period is not possible, as patients need to be constantly monitored to ensure effective treatment, thus preventing thromboembolic events. The study was conducted for twelve months, as follows:

1. Patients received a kit with a Coagulometer-CoaguChek® (Roche Diagnostics, Switzerland) and the necessary test strips for use during the period established, as well as written instructions on how to take the measurements, and were registered on the monitoring platform.
2. Patients received periodic text messages on their smartphones to report the INR value, and they responded to messages regarding their symptoms related to anticoagulant therapy and the INR value.
3. The clinical team received notifications if patients' reports had been assessed outside therapeutic standards and then sent a text message back with the medication adjustment.

ELIGIBILITY:
Inclusion Criteria:

* equal or more than 18 years old and with a smartphone

Exclusion Criteria:

* analphabetism, poor health, low digital literacy level and inability to use the RPM alone or with caregiver support

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-10-10 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Time in Therapeutic Range (TTR) for International Normalized Ratio (INR) | From enrollment to the end of treatment at 12 months
  The primary endpoint was the patient's TTR for INR values among the programs, i.e., a comparison between SOC and RPM over time. The TTR for INR value was self-measured by the portable monitor and calculated by the Rosendaal method of lineal interpolation

SECONDARY OUTCOMES:
Number of events of hypocoagulation symptoms | From enrollment to the end of treatment at 12 months
  Zero is equivalent to no hypoagulation symptoms and more than one indicates a symptom
Patient Experience and Satisfaction | From enrollment to the end of treatment at 12 months
  . A questionnaire with 13 self-reported questions was used to evaluate patient experience and satisfaction. The first four questions measured experience, while the following nine focused on satisfaction. The responses were rated on a scale of disagree to agree, with 1-4 points assigned to each response. To prevent ceiling and floor effects in our tool, the questions numbered '2', '11', and '12' were calculated as "inverted," and an optional open question was included. The questionnaire used to assess experience and satisfaction is not validated, precluding external validity. Still, it was used due to the lack of instruments in Portuguese language to assess the experience and satisfaction of digital health RPM-based systems.
Costs | From enrollment to the end of treatment at 12 months
  The method used in the trial compared the average cost per patient in standard of care (SOC) versus remote patient monitoring (RPM) using the Time-Driven Activity-Based Costing (TDABC) method from the perspective of the Public National Healthcare Service (NHS). The method involved mapping patient pathway activities and identifying direct costs such as healthcare professionals, facilities, equipment and technology, and consumables. Costs for healthcare professionals, equipment and technology, and facilities were determined based on market value, depreciation rate, and public salary scale. Travel costs for patients undergoing SOC were considered, and all monetary values are in Euros as of 2023.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Rita Londral, PhD, Principal Investigator — Value for Health CoLAB
Locations (1):
- Hospital de Santa Marta, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sharma P, Scotland G, Cruickshank M, Tassie E, Fraser C, Burton C, Croal B, Ramsay CR, Brazzelli M. Is self-monitoring an effective option for people receiving long-term vitamin K antagonist therapy? A systematic review and economic evaluation. BMJ Open. 2015 Jun 25;5(6):e007758. doi: 10.1136/bmjopen-2015-007758. PMID 26112222
- [Background] Menendez-Jandula B, Garcia-Erce JA, Zazo C, Larrad-Mur L. Long-term effectiveness and safety of self-management of oral anticoagulants in real-world settings. BMC Cardiovasc Disord. 2019 Aug 2;19(1):186. doi: 10.1186/s12872-019-1168-2. PMID 31375070
- [Background] Azevedo S, Guede-Fernandez F, von Hafe F, Dias P, Lopes I, Cardoso N, Coelho P, Santos J, Fragata J, Vital C, Semedo H, Gualdino A, Londral A. Scaling-up digital follow-up care services: collaborative development and implementation of Remote Patient Monitoring pilot initiatives to increase access to follow-up care. Front Digit Health. 2022 Dec 7;4:1006447. doi: 10.3389/fdgth.2022.1006447. eCollection 2022. PMID 36569802
- [Background] Wu Y, Wang X, Zhou M, Huang Z, Liu L, Cong L. Application of eHealth Tools in Anticoagulation Management After Cardiac Valve Replacement: Scoping Review Coupled With Bibliometric Analysis. JMIR Mhealth Uhealth. 2024 Jan 5;12:e48716. doi: 10.2196/48716. PMID 38180783
- [Background] Huang Y, Xie Y, Huang L, Han Z. The Value of Anticoagulation Management Combining Telemedicine and Self-Testing in Cardiovascular Diseases: A Meta-Analysis of Randomized Controlled Trials. Ther Clin Risk Manag. 2023 Mar 14;19:279-290. doi: 10.2147/TCRM.S395578. eCollection 2023. PMID 36941980
- [Derived] Guede-Fernandez F, Silva Pinto T, Semedo H, Vital C, Coelho P, Oliosi ME, Azevedo S, Dias P, Londral A. Enhancing postoperative anticoagulation therapy with remote patient monitoring: A pilot crossover trial study to evaluate portable coagulometers and chatbots in cardiac surgery follow-up. Digit Health. 2024 Aug 6;10:20552076241269515. doi: 10.1177/20552076241269515. eCollection 2024 Jan-Dec. PMID 39139188